CLINICAL TRIAL: NCT04686799
Title: Evaluating the Feasibility of Subantimicrobial-dose Doxycycline for Elbow Tendinopathy
Brief Title: Doxycycline for Elbow Tendinopathy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-1582
Record Dates: First submitted 2020-11-06; First posted 2020-12-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-01

CONDITIONS: Lateral Epicondylitis; Lateral Epicondylitis, Left Elbow; Lateral Epicondylitis, Right Elbow; Lateral Epicondylitis, Unspecified Elbow; Lateral Epicondylitis (Tennis Elbow) Bilateral; Medial Epicondylitis; Medial Epicondylitis, Right Elbow; Medial Epicondylitis, Left Elbow
Keywords: Feasibility; efficacy
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: The plan for achieving the specific aims is to first assess patient receptiveness by screening patients with symptomatic lateral or medial elbow tendinopathy for eligibility and tracking the proportion of eligible patients who decline participation in the study due to not wanting to take an extended course of SD-doxycycline. 25 subjects will given SD-doxycycline and have the tendinopathy grade measured by ultrasound. The medication will be prescribed for 12 weeks during which time logs will be used to track compliance and monitor side effects. This will be done in combination with usual care, which includes a home exercise program, a counterforce brace, and over-the-counter pain medication to use as needed. Clinical effectiveness outcomes will include patient reported outcomes, ultrasound tendinopathy grade, grip strength, and markers of MMP activity and collagen production/connective tissue anabolism.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SD-doxycycline group (Experimental): 12 weeks SD-doxycycline: doxycycline hyclate 20 mg tablet by mouth twice daily
  Interventions: Drug: Doxycycline Hyclate 20 MG

INTERVENTIONS:
Drug: Doxycycline Hyclate 20 MG — Subjects will receive doxycycline 20 mg BID

SUMMARY:
To evaluate the feasibility of subantimicrobial -dose (SD) doxycycline to improve outcomes of nonsurgical management of elbow tendinopathy via matrix metalloproteinase (MMP) inhibition as well as evaluate if participants will be compliant to with prescribed medication and exercise treatment. Our working hypothesis is that patients with elbow tendinopathy will be receptive to treatment with SD-doxycycline and compliant with the prescribed treatment.

DETAILED DESCRIPTION:
: elbow tendinopathy is a common condition among athletes and the general population. It can result in significant disability and time loss from work. Despite traditional nonsurgical treatment, symptoms often persist for more than 6 months. Second-line treatments, such as platelet rich plasma injections and extracorporeal shock wave therapy, have limited evidence and are often cost-prohibitive. There remains a need for additional cost-effective nonsurgical treatment for elbow tendinopathy.

Purpose: To evaluate the feasibility of subantimicrobial -dose (SD) doxycycline to improve outcomes of nonsurgical management of elbow tendinopathy via matrix metalloproteinase (MMP) inhibition as well as evaluate if participants will be compliant to with prescribed medication and exercise treatment. Our working hypothesis is that patients with elbow tendinopathy will be receptive to treatment with SD-doxycycline and compliant with the prescribed treatment.

Methods: This study will enroll 25 otherwise healthy males and females ages 18 and up with ≥ 6 weeks of symptomatic lateral or medial elbow tendinopathy. Subjects will receive doxycycline 20 mg BID (twice a day) for 12 weeks. Usual care will also be provided with a home exercise program and a counterforce brace. The proportion of eligible patients who elect to participate in the study will be tracked as a measure of receptiveness. Biweekly logs will be collected to monitor for treatment side effects and track compliance. Patient reported outcomes will include quick Disabilities of the Arm Shoulder and Hand score (qDASH) and Patient-Rated Tennis Elbow Evaluation (PRTEE) at baseline, 4, 8, and 12 weeks. Ultrasound tendinopathy grade and grip strength will be measured at baseline and 12 weeks. Blood will be drawn to assess MMP activity and collagen production/connective tissue anabolism at baseline and 12 weeks.

Significance: This study will provide the necessary data to design a phase two-a trial of a safe, low-cost adjuvant treatment for a common condition treated by sports medicine and primary care physicians. If found to be beneficial for elbow tendinopathy, SD-doxycycline may have utility in other types of tendinopathy as well.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages of 18 and up
* Atraumatic unilateral elbow pain of ≥ 6 weeks duration
* Diagnosed clinically as lateral or medial elbow tendinopathy
* Activity-related lateral or medial elbow pain
* Tenderness of the lateral or medial epicondyle
* Pain with gripping and/or resisted wrist extension with the elbow extended
* Pain with passive wrist flexion and finger with the elbow extended
* Internet access to complete electronic surveys

Exclusion Criteria:

* Prior surgery of the affected elbow
* Prior injection of the affected lateral or medial epicondyle or extensor tendons
* Prior extracorporeal shockwave therapy to the affected elbow
* Suspicion for radial tunnel syndrome (tenderness distal to the lateral epicondyle in the area of the supinator muscle dorsally, pain with resisted supination with the elbow extended, and/or weakness of the extensor digitorum communis)
* Separate upper extremity injury or condition that would interfere with full participation in the home exercise program
* Fluoroquinolone-associated tendinopathy
* Ligamentous laxity on exam
* Evidence of osteoarthritis or osteochondral lesion on radiographs
* Autoimmune condition
* Pregnant, intend to become pregnant, or breastfeeding
* Premenopausal women who are not using contraception
* Allergy to doxycycline or other tetracyclines
* Current esophagitis or peptic ulcer disease
* Current use of medication for which there is a drug interaction with doxycycline
* Who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primarily a feasibility study of SD-doxycycline as an adjunctive treatment for elbow tendinopathy (Compliance) | 12 weeks
  Compliance: At the end of the study, compliance will be calculated using the number of self-reported doses taken divided by the number of prescribed doses (twice daily x 7 days per week x 12 weeks = 168 doses).
Receptiveness | 12 weeks
  The number of patients who enroll in study divided by the number eligible patients minus the number of patients who decline due to reasons unrelated to the prescribed treatment, e.g., unable to return for second study visit. This will be measured at time of study recruitment.

SECONDARY OUTCOMES:
Clinical outcomes - qDASH | 12 weeks
  quick Disabilities of the Arm Shoulder and Hand score (by qDASH score) at baseline, 4, 8, and 12 weeks
Clinical outcomes - PRTEE | 12 weeks
  Patient-Rated Tennis Elbow Evaluation (by PRTEE test ) at baseline, 4, 8, and 12 weeks
Secondarily, clinical outcomes will be measured to provide preliminary data to power a future randomized controlled trial. (Ultrasound tendinopathy grade) | 12 weeks
  Ultrasound tendinopathy grade at baseline at 12 weeks - by ultrasound
Clinical outcomes - Grip strength | 12 weeks
  Grip strength at baseline and 12 weeks - measure by hand-held dynamometer
Clinical outcomes - MMP | 12 weeks
  Matrix metalloproteinase (MMP) inhibition activity and collagen production/connective tissue anabolism at baseline and 12 weeks - measure by blood test

CONTACTS AND LOCATIONS:
Overall Officials: Brett G Toresdahl, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following study publication. No end date.
Access Criteria: Any purpose